CLINICAL TRIAL: NCT03923140
Title: Efficacy and Safety of Tranilast in Patients With Cryopyrin-Associated Periodic Syndrome (CAPS): A Single-Arm Prospective Cohort Study
Brief Title: A Clinical Study of Tranilast in the Treatment of Cryopyrin-Associated Periodic Syndrome (CAPS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Hongmei Song, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-1921
Record Dates: First submitted 2019-04-14; First posted 2019-04-22 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Cryopyrin-Associated Periodic Syndromes
Keywords: Cryopyrin-Associated Periodic Syndromes; Tranilast; Efficacy; Safety
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — tranilast

STUDY DESIGN:
Intervention Model Description: a single-arm prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tranilast (Experimental): 5mg/kg.d for juvenile patients with a maximum dose of 0.3g per day; 0.1g each time, three times a day for adults patients
  Interventions: Drug: Tranilast

INTERVENTIONS:
Drug: Tranilast — 5mg/kg.d for juvenile patients with a maximum dose of 0.3g per day; 0.1g each time, three times a day for adults patients
  Other Names: Rizaben

SUMMARY:
This is a prospective cohort study to observe the efficacy and safety of tranilast in CAPS patients. The investigators would analyze the changes in Auto-Inflammatory Diseases Activity Index (AIDAI) before and after treatment as well as changes in inflammatory markers, patients' and physician's global assessment of disease activity to determine the efficacy and safety of tranilast.

DETAILED DESCRIPTION:
Seventy-one patients with CAPS will be recruited. After signing the informed consent, they will be administrated with tranilast (For juvenile patients, 5mg/kg.d with a maximum dose of 0.3g per day; For adult patients, the dose is 0.1g each time, three times a day). These patients will be followed up for 6 months. AIDAI is recorded by patients' or their parents one month before the start of treatment, and at the 1st, 3rd and 6th month after the treatment. Inflammatory markers, and patients' and physician's global assessment of disease activity will be assessed during the 1st, 3rd and 6th month follow-up. Side effects will be monitored and recorded as well. Experimental data before and after the administration of tranilast will be analyzed and be statistically processed, to figure out whether tranilast is effective and safe for CAPS patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following diagnostic criteria of CAPS and have pathogenic mutation(s) in NLRP3 gene.

  1. Raised inflammatory markers (CRP/SAA) (mandatory criteria)
  2. ≥2 of 6 CAPS typical signs/symptoms:

     1. Urticaria-like rash;
     2. Cold/stress triggered episodes;
     3. Sensorineural hearing loss;
     4. Musculoskeletal symptoms (arthralgia/arthritis/myalgia);
     5. Chronic aseptic meningitis;
     6. Skeletal abnormalities (epiphyseal overgrowth/frontal bossing).

Exclusion Criteria:

* Patients will not be included if meets any of the following criteria:

  1. Being treated with IL-1 inhibitor, other biological agents and immunosuppressants
  2. Pregnant and lactating women
  3. Serious organ function failure, expected life time less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Auto-Inflammatory Diseases Activity Index score after 6-month treatment over baseline | The previous 1 month before treatment and the 6th month after treatment
  Patients or their parents completed a 1-month (31 days) prospective diary with 12 yes/no items( Fever ≥38°C, Overall symptoms, Abdominal pain, Nausea/vomiting, Diarrhoea, Headaches, Chest pain, Painful nodes, Arthralgia or myalgia, Swelling of the joints, Eye manifestations, Skin rash) at the previous 1 month before treatment, and the 6th month after treatment . Each item of this diary was dichotomised as no (0)=absence of symptom or yes (1)=presence of symptom. The calculation of the Auto-Inflammatory Diseases Activity Index score is straightforward, consisting of the sum of all 12 items (0-372 in a month of 31 days). Higher values represent higher disease activity.

SECONDARY OUTCOMES:
Changes in Auto-Inflammatory Diseases Activity Index score at the 1st and 3rd month over baseline | The previous 1 month before treatment and the 1st and 3rd month after treatment
  Patients or their parents completed a 1-month (31 days) prospective diary with 12 yes/no items( Fever ≥38°C, Overall symptoms, Abdominal pain, Nausea/vomiting, Diarrhoea, Headaches, Chest pain, Painful nodes, Arthralgia or myalgia, Swelling of the joints, Eye manifestations, Skin rash) at the previous 1 month before treatment, and the 1st and 3rd month after treatment . Each item of this diary was dichotomised as no (0)=absence of symptom or yes (1)=presence of symptom. The calculation of the Auto-Inflammatory Diseases Activity Index score is straightforward, consisting of the sum of all 12 items (0-372 in a month of 31 days). Higher values represent higher disease activity.
Changes in inflammatory markers, including C-reactin protein, erythrocyte sedimentation rate, serum amyloid protein, interleukin-1β and interleukin-18， at 1, 3 and 6 months over baseline | Baseline and at 1, 3 and 6 months after treatment
  C-reactin protein, erythrocyte sedimentation rate, serum amyloid protein, interleukin-1β and interleukin-18 are measured at baseline，1, 3 and 6 months after treatment.
Changes in physician global assessment of disease activity on a 0-10 visual analog scale (VAS) at 1, 3 and 6 months over baseline | Baseline and 1, 3 and 6 months after treatment
  Visual analogue scale (VAS) for overall disease activity were completed by the physician at each visit (Baseline and 1, 3 and 6 months after treatment).
Changes in parent/patient global assessment of well-being on a 0-10 visual analogue score (VAS) at 1, 3 and 6 months over baseline | Baseline and 1, 3 and 6 months after treatment
  Visual analogue scale (VAS) for overall disease activity were completed by the parent/patient at each visit (Baseline and 1, 3 and 6 months after treatment).
Changes in CSF white blood cell count for CINCA patients | Baseline and 6 months after treatment.
  For CINCA patients, Lumbar punctures (LPs) were performed at baseline and 6 months after treatment.
Changes in MRI of the brain and inner ear for CINCA patients | Baseline and 6 months after treatment.
  For CINCA patients, MRIs with gadoliniumenhanced fluid-attenuated inversion recovery (FLAIR) sequences of the brain and inner ear were performed and scored at baseline and 6 months after treatment.
Changes in audiology data for CINCA patients | Baseline and 6 months after treatment.
  For CINCA patients, Hearing assessment included audiological evaluations. Outcomes in each ear were categorised as 'stable' or 'worsened', according to a modification of the American Speech and Hearing Association (ASHA) criteria, comparing the results at 6 months after treatment over baseline.
Number of participants with adverse effect | Up to 6 months
  Treatment-related adverse effect, including abnormal liver function, hematuria and decreased white blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Song, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No